CLINICAL TRIAL: NCT07160673
Title: Tech-based Respite Care for Caregivers and Homebound Older Adults: A Randomized Controlled Trial
Brief Title: Tech-based Respite Care for Caregivers and Homebound Older Adults
Acronym: TechRespiteRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong University (Other)
Responsible Party: Principal Investigator, Linda Dong-Ling Wang, Research Assistant Professor, Hong Kong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0048-007
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Caregiver Stress; Social Isolation in Older Adults; Cognitive Decline in Older Adults; Depression in Older Adults; Anxiety in Older Adults
Keywords: Virtual Reality; Respite Care; Caregivers; Older Adults; Randomized Controlled Trial; Mental Health; Cognitive Function; uality of Life
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR Intervention Group (Experimental): Caregivers and homebound older adults will receive 4 weeks of VR-based respite sessions.
  Interventions: Device: VR-based Respite
- Video Control Group (Active Comparator): Caregivers and homebound older adults will receive 4 weeks of video-based respite sessions.
  Interventions: Device: Video-based Respite
- Usual Care Group (No Intervention): Caregivers and homebound older adults will receive no additional intervention.

INTERVENTIONS:
Device: VR-based Respite — Caregivers and homebound older adults will receive 4 weeks of VR-based respite sessions. 4 weeks (1 session/week; 30 min/session) of immersive VR sessions using SilVR Adventures platform. Sessions include virtual travel destinations (e.g., cities, natural wonders) and social activities (e.g., group tours). Facilitated by trained research staff, with 5-10 minutes viewing and 20 minutes reflection/discussion.
  Arms: VR Intervention Group
Device: Video-based Respite — Caregivers and homebound older adults will receive 4 weeks of video-based respite sessions. 4 weeks (1 session/week; 30 min/session) of non-immersive video sessions with content similar to VR themes (e.g., landscapes, cultural events). Facilitated by trained research staff, with post-video discussion. EEG data collected during viewing to assess emotional states.
  Arms: Video Control Group

SUMMARY:
The goal of this study is to examine the effectiveness of VR-based respite in improving cognitive function, mental health, and quality of life in caregivers and homebound older adults compared to a control group using videos and a usual care group. Participants are randomly assigned to one of three groups: VR intervention, video control, or usual care.

The VR group receives immersive VR sessions using the SilVR Adventures platform. The video group receives non-immersive video sessions with similar content. The usual care group receives no additional intervention.

Assessments are conducted at baseline, immediate post-intervention, and 3 months post-intervention to measure changes in depression, anxiety, loneliness, quality of life, and other outcomes. The intervention dosage will be 4 weeks (1 sessions/week; 30 min/session).

Secondarily, the study explores differences in effectiveness between caregivers and homebound older adults, and potential moderators or mediators such as baseline health status, technological literacy, and social support.

DETAILED DESCRIPTION:
All participants will provide informed consent at the time of enrolment. Both caregivers (CGs) and care recipients (CRs) will complete assessments at baseline.

CRs are assessed for cognitive function (using Mini-Mental State Examination - MMSE) and other health indicators. CGs are assessed for mental health, quality of life, and caregiving burden.

Participants are randomized into three groups: VR intervention (n=30 dyads), video control (n=30 dyads), or usual care (n=30 dyads). Randomization is stratified by CG age (<60 vs. ≥60) and CR cognitive status (MMSE <24 vs. ≥24).

As the intervention, the VR group receives 4 weekly 30-minute sessions of immersive VR experiences (e.g., virtual travel and social activities) facilitated by trained research staff. The video group receives 4 weekly 30-minute sessions of non-immersive videos with similar themes, also facilitated. The usual care group receives no additional intervention beyond community services.

At the end of the intervention, participants complete assessments again to measure changes in physical and mental health.

All participants will be contacted for follow-up assessment 3 months after the completion of intervention.

ELIGIBILITY:
Caregivers (CGs)

Inclusion Criteria:

* Aged 18 or above
* Provide care to at least one homebound older adult (aged 60 or above)
* Provide no less than 6 hours of caregiving per week
* Able to communicate in either Cantonese, Mandarin or English
* Willing to participate for the entire duration
* Able to tolerate VR headset for at least 5 minutes (no severe motion sickness/epilepsy)

Exclusion Criteria:

* History of severe psychiatric disorders (e.g., schizophrenia, bipolar)
* Severe cognitive impairment (MMSE <10)
* Major neurological diseases (e.g., recent stroke, severe Parkinson's)
* Uncorrectable visual/hearing impairments affecting VR/video
* Unable to tolerate VR due to motion sickness or discomfort
* Care recipient receiving long-term care service that conflicts with study

Care Recipients (CRs)

Inclusion Criteria:

* Aged 60 or above
* Homebound (unable to leave home without assistance)
* Stable medical condition
* Willing to participate for the entire duration
* Able to tolerate VR headset for at least 5 minutes (no VR contraindications)
* Able to understand and provide informed consent Exclusion Criteria: Same as CGs, plus MMSE <10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depression and anxiety on PHQ-4 after intervention | Baseline, Immediate after intervention, and 3 months after intervention
  The Patient Health Questionnaire-4 (PHQ-4) is a validated 4-item scale measuring depression and anxiety over the past two weeks. Rated on a 4-point scale from "not at all" to "nearly every day."
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in quality of life on EQ-5D-5L after intervention | Baseline, Immediate after intervention, and 3 months after intervention
  EQ-5D-5L is a validated 6-item scale measuring quality of life across 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) plus a visual analogue scale (EQ-VAS, 0-100). Higher scores indicate better quality of life.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in loneliness on UCLA Loneliness Scale after intervention | Baseline, Immediate after intervention, and 3 months after intervention
  The 3-item UCLA Loneliness Scale is a validated tool measuring feelings of loneliness and social isolation. The total score can range from 3 to 9. Higher scores indicate greater degrees of loneliness.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in subjective happiness on Subjective Happiness Scale after intervention | Baseline, Immediate after intervention, and 3 months after intervention
  The Subjective Happiness Scale is a validated 4-item scale measuring global subjective happiness on a 7-point Likert scale. Reverse the score for Item 4. Calculate the mean of all four item scores (the three regular scores plus the reversed score from Item 4). The total score ranges from 1 to 7. Higher scores indicate greater subjective happiness.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)

SECONDARY OUTCOMES:
Change from baseline in cognitive function on MMSE after intervention (For CRs only) | : Baseline, Immediate after intervention, and 3 months after intervention
  The Mini-Mental State Examination (MMSE) is a validated 30-point questionnaire assessing cognitive function (orientation, memory, attention, etc.). Scores range from 0-30; higher scores indicate better function.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in role captivity on Pearlin's model after intervention(For CGs only) | Baseline, Immediate after intervention, and 3 months after intervention
  Pearlin's Role Captivity Scale is a 3-item tool measuring internal strain of caregiving role on a 4-point Likert scale. The total scores range from 3 to 12. Higher scores indicate greater role captivity.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in technology acceptance on STAM after intervention | Baseline and Immediate after intervention
  The Senior Technology Acceptance Model (STAM) is a validated 14-item scale consisted of a 4-factor structure (Attitudinal beliefs, Control beliefs, Gerontechnology anxiety, and Health). Each construct is measured by several items on a 10-point scale. For each of the four factors, calculate a composite score. This is done by taking the mean of all the items that load onto that factor. Additionally, a higher global score indicates a more positive overall attitude towards technology acceptance.
  Change = Immediate after intervention - baseline
4. Change from baseline in quality of life on OPQOL-brief after intervention (For CRs only) | Baseline, Immediate after intervention, and 3 months after intervention
  The Older People's Quality of Life - brief questionnaire (OPQOL-brief) is a validated 13-item scale measuring QoL domains (health, social relationships, independence) on a 5-point Likert scale. Add together the scores from all 13 items after the reverse-scoring has been completed. The total score ranges from 13 to 65. A higher total score indicates a better self-reported quality of life.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)
Change from baseline in caregiving burden on CZBI-short after intervention (For CGs only) | Baseline, Immediate after intervention, and 3 months after intervention
  The Cantonese short version of the Zarit Burden Interview (CZBI-short) is a validated 12-item scale measuring caregiver burden on a 5-point Likert scale (0=never to 4=very frequently). Scores range from 0-48; higher scores indicate greater burden.
  Change = (Immediate after intervention - baseline) and (3 months after intervention - baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Sau Po Centre on Ageing, HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No